CLINICAL TRIAL: NCT07386223
Title: HEAL-FHA: Health and Lifestyle Support for Functional Hypothalamic Amenorrhea
Brief Title: Health and Lifestyle Support for Functional Hypothalamic Amenorrhea
Acronym: HEAL-FHA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); FoU Centrum, Landstinget Sörmland (Other Government)
Responsible Party: Principal Investigator, Hedvig Engberg, Assistant Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-05586-01
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Hypothalamic Amenorrhea, Functional
Keywords: psychoeduction; lifestyle change; menstrual restoration; amenorrhea
MeSH Terms: conditions — Amenorrhea | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducational Intervention (Experimental): Participants in this arm will take part in a 10-week psychoeducational health and lifestyle program designed to support behavioural change related to recovery from Functional Hypothalamic Amenorrhea (FHA). The intervention includes weekly modules focusing on nutrition, exercise behaviours, stress management, and recovery-promoting habits, delivered with evidence-based educational content and practical exercises. Participants will also complete questionnaires and provide blood samples at scheduled timepoints and will be followed for 9 months after the intervention.
  Interventions: Behavioral: Psychoeducaction or treatment as usual
- Treatment as Usual (TAU) (Active Comparator): Participants in this arm will receive treatment as usual for Functional Hypothalamic Amenorrhea, which may include general clinical advice, routine follow-up, and standard information provided by healthcare services. No structured psychoeducational program will be offered. Participants will complete questionnaires and provide blood samples at the same timepoints as the intervention group.
  Interventions: Other: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Psychoeducaction or treatment as usual — 10 week psychoeducaction or treatment as usual
  Arms: Psychoeducational Intervention
Other: Treatment as usual (TAU) — Standard FHA management provided in routine clinical care.
  Other Names: Standard FHA management provided in routine clinical care.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The goal of this clinical trial is to learn whether a 10-week psychoeducational health and lifestyle intervention can help women with Functional Hypothalamic Amenorrhea (FHA) restore their endocrine balance and menstrual cycles.

The main questions the study aims to answer are:

Does the intervention lead to the return of regular menstrual bleeding? Does it improve hormonal markers associated with FHA recovery? To answer these questions, researchers will compare the 10-week psychoeducational intervention with treatment as usual (TAU). This comparison will help determine whether the structured program leads to faster or more reliable recovery of menstrual and endocrine function than the care women typically receive today.

Participants will:

Take part in a 10-week psychoeducational program focusing on health behaviors important for FHA recovery (intervention group) or receive treatment as usual (comparison group) Complete questionnaires and health assessments Provide blood samples to measure hormone levels Take part in a gynecological exam to monitor ovary activity and endometrial thickness Be followed for 9 months after the program to track progress This study builds on a previous feasibility study and will help determine whether the intervention is effective and should be used more widely to support women with FHA.

DETAILED DESCRIPTION:
The study a randomized, controlled, multicentre trial evaluating a 10-week psychoeducational health and lifestyle intervention with a 9-month follow-up period in women with Functional Hypothalamic Amenorrhea (FHA).

Background and Significance FHA is a functional endocrine condition that can be reversed through behavioural and lifestyle changes. A structured psychoeducational program may support these changes by improving knowledge, motivation, and self-management skills. The intervention will be compared with treatment as usual (TAU) to determine whether it leads to superior restoration of menstrual and endocrine function.

Study Aim The aim of this study is to evaluate whether a 10-week psychoeducational intervention is effective in restoring menstrual and endocrine function in women with FHA.

Study Setting and Participants A total of 70 women with FHA will be recruited following the same procedures used in Study 1. Participants who meet inclusion criteria and provide informed consent will enter the trial. Those who meet exclusion criteria will receive appropriate clinical information, standard care, or referral to relevant healthcare services.

Power Analysis The sample size calculation is based on findings from a previous trial evaluating an individualized Cognitive Behavioural Therapy (CBT) intervention, where ovarian recovery occurred in 87.5% of participants receiving CBT compared with 33% in the observation group. For the current trial, the psychoeducational intervention is expected to yield a slightly lower effect (estimated 70% recovery). With 80% power and α = 0.05, 28 participants per group are required to detect this difference. Allowing for up to 15% attrition, the study will recruit 35 participants per arm.

Study Design The study uses a two-arm, parallel-group, superiority randomized controlled design with 1:1 allocation. Randomization will be conducted by Karolinska Trial Alliance (KTA). Participants will undergo baseline psychiatric screening with MINI+ and complete validated psychological questionnaires at baseline, post-treatment, and at 9-month follow-up. These assessments will capture stress, coping, symptoms of anxiety and depression, eating disorder symptoms, exercise behaviours, and personality traits associated with FHA. Hormonal analyses will be performed at baseline, post-treatment, and at 3-, 6-, and 9-month follow-up.

Data and Sample Collection The qualitative and quantitative findings from the feasibility study will inform refinement of the final study protocol. All questionnaire data will be collected electronically via REDCap. Hormonal analyses will include repeated measures of LH and additional hormones related to ovarian function. Participants will report all episodes of vaginal bleeding or spotting during the study period. If bleeding occurs, estradiol and progesterone will be measured 21 days later to assess for ovulation.

Outcome Measures The primary outcome is restoration of menstrual function. Secondary outcomes include normalization of luteinizing hormone (LH; reference range 2.4-13 IU/L) as a marker of restored GnRH pulsatility, as well as reductions in self-reported mental health symptoms at 9-month follow-up. Negative effects will be monitored using self-report instruments.

Statistical Analysis Primary treatment response is defined as restoration of menstruation; secondary response is defined as normalization of LH levels. Planned analyses include hypothesis testing of pre-/post-treatment changes using two-sided paired t-tests. Additional analyses will follow a predefined statistical analysis plan.

Ethical Considerations Informed consent will be obtained from all participants. Studies are approved by the Swedish Ethical Review Authority (Dnr 2023-05586-01). An amendment for Study 2 is planned. Participants will complete questionnaires, provide blood samples, and undergo a gynecological examination. The overall risk to participants is considered low, and adverse events will be monitored throughout the study period.

ELIGIBILITY:
Inclusion Criteria

* female
* aged 18-42 years
* fulfill criteria for diagnosis of functional hypothalamic amenorrhea (hypogonadotropic hypogonadism)
* basic proficiency in Swedish
* access to a computer.

Exclusion Criteria:

* Lack of proficiency in language
* evere psychiatric co-morbidity e.g. psychosis or active eating disorders (anorexia nervosa).

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with return of spontaneous menstrual bleeding within 9 months | Restoration of menstruation after 9 months of follow-up
  Restoration of menstruation is defined as a spontaneous menstrual bleed observed reported by the participants. Hormonal assessment will occur on cycle day 21 of the next menstrual cycle following intervention. The outcome will be reported as the number and proportion of participants who experience menstrual restoration.
Change in serum FSH, LH, and estradiol | 12 months
  For participants who have not experienced menstruation during follow-up serum FSH, LH, and estradiol levels will be measured to evaluate hormonal improvement. Changes from baseline will be reported as mean ± SD and as the proportion of participants showing increase in estradiol consistent with improved ovarian function.

CONTACTS AND LOCATIONS:
Locations (1):
- Kvinnohälsan Karolinska Universitetssjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
What data will be shared:
  De-identified individual participant data collected during the trial, including:
  Demographics (age, sex) Clinical assessments and questionnaire responses Hormonal measurements (LH, estradiol, progesterone) Menstrual cycle and ovulation data Psychological and behavioral assessments
  Other documents to be shared:
  Data dictionary describing all variables and coding used Study protocol and statistical analysis plan
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When data will become available and for how long:
  Data will be available 6 months after publication of the primary trial results and will remain accessible for 5 years.
Access Criteria: By what access criteria:
  Data will be available to qualified researchers for scientific purposes following submission of a research proposal and approval by the trial steering committee. Requests should be sent to the corresponding author or data custodian (contact information provided in the study publication).Data will be shared via a secure data repository